CLINICAL TRIAL: NCT04268628
Title: Exploratory Evaluation of Genetic Polymorphism and Pharmacodynamic Parameters in Samples of Abira-DES Study Subjects (NCT02217566) - Subjects With Metastatic Castration-Resistant Prostate Cancer Treated With Abiraterone Acetate Following Unresponsive Treatment With Diethylstilbestrol.
Brief Title: A Study of Pharmacodynamic and Genetic Parameters of Abira-DES Study Participants (NCT02217566) - Participants With Metastatic Castration-Resistant Prostate Cancer Treated With Abiraterone Acetate Following Unresponsive Treatment With Diethylstilbestrol
Acronym: EXPLORE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108736; 212082PCR0026 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Participants with mCRPC: Participants with metastatic castration resistant prostate cancer (mCRPC) will be evaluated for genetic polymorphism and pharmacodynamic parameters from serum and plasma samples collected during the Abira-DES study (NCT02217566). Serum and plasma samples were collected after use of diethylstilbestrol (DES) and subsequent abiraterone acetate therapy. Peripheral blood samples were collected prior to initiation of abiraterone acetate therapy, after 12 weeks of therapy, and at the time of disease progression (evaluated by prostate specific antigen [PSA] response).
  Interventions: Other: Serum and plasma samples analysis

INTERVENTIONS:
Other: Serum and plasma samples analysis — This is a non-interventional study and no drug will be given as part of this study. Serum and plasma samples will be collected from the participants with metastatic castration-resistant prostate cancer to evaluate genetic polymorphism and pharmacodynamic parameters.

SUMMARY:
The primary purpose of this study is to evaluate the influence of HSD3B1 (1245C) germline variant and potential pharmacodynamic markers on abiraterone activity in participants with metastatic castration-resistant prostate cancer after unresponsive use of diethylstilbestrol.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of prostate adenocarcinoma without neuroendocrine or small cell differentiation and was a participant in the Abira-DES study (NCT0221756), which includes: diethylstilbestrol pretreatment for castration-resistant prostate cancer with evidence of disease progression or grade 3/4 toxicity with diethylstilbestrol; metastatic disease confirmed by bone examination or metastatic lesions by computed tomography or magnetic resonance
* Abiraterone acetate therapy during the Abira-DES study (NCT0221756), and peripheral blood samples have been collected from at least of the three proposed study timepoints
* Must sign, and/or his/her legally acceptable representatives, where applicable, must sign the ICF allowing the use of clinical data and biological samples in accordance with local requirements. For deceased participants who did not provide consent prior to death, permission to research their information must meet local requirements

Exclusion Criteria:

- Having withdrawn the consent to use the samples collected during their participation in the Abira-DES study (NCT02217566)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study comprised of participants with metastatic castration-resistant prostate cancer with disease progression following the use of diethylstilbestrol (DES) who participated in the Abira-DES study (NCT02217566) in which they were treated with abiraterone acetate.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with and Without HSD3B1 (1245C) Germline Variant' | Up to 12 months
  Percentage of participants with and without HSD3B1 (1245C) germline variant will be determined to evaluate the influence of HSD3B1 (1245C) germline variant on the response to abiraterone as a predictive fact.

SECONDARY OUTCOMES:
Levels of HSD3B1 (1245C) Germ Variant | Up to 12 months
  Levels of HSD3B1 (1245C) germline variant will be determined to evaluate the response to abiraterone acetate as a predictive factor.
Levels of Metabolite Delta-(4)-Abiraterone (D4A) During the Abiraterone Acetate During Treatment Phase | 12 Weeks
  Levels of metabolite D4A during the abiraterone acetate during treatment phase will be evaluated.
Testosterone Levels in Participants Treated with Abiraterone Acetate | Up to 12 months
  Testosterone levels of participants treated with abiraterone acetate will be evaluated by the molecular analyses.
SDHEA Levels in Participants Treated with Abiraterone Acetate | Up to 12 months
  SDHEA levels of participants treated with abiraterone acetate will be evaluated by the molecular analyses.
Correlation Between HSD3B1 (1245C) Variant and Testosterone Levels | Up to 12 months
  Correlation between HSD3B1 (1245C) variant and testosterone levels will be reported. The genotyping of the HSD3B1 (1245 A> C) germline variant will be performed by Sanger sequencing.
Correlation Between HSD3B1 (1245C) Variant and SDHEA Levels | Up to 12 months
  Correlation between HSD3B1 (1245C) variant and SDHEA levels will be reported. The genotyping of the HSD3B1 (1245 A> C) germline variant will be performed by Sanger sequencing.
Correlation Between HSD3B1 (1245C) Variant and Clinical Response | Up to 12 months
  Correlation between HSD3B1 (1245C) variant and clinical response will be performed by univariate and multivariate analyses.
Correlation Between D4A Levels with Testosterone Dosage | Up to 12 months
  Testosterone ultrasensitive dosages will be performed on participant serum samples. Testosterone dosage will be performed by liquid chromatography coupled with tandem mass spectrometry.
Correlation Between D4A Levels with SDHEA Dosage | Up to 12 months
  SDHEA ultrasensitive dosages will be performed on participant serum samples. Dosage will be performed by liquid chromatography coupled with tandem mass spectrometry.
Correlation Between D4A Levels with Clinical Response | Up to 12 months
  Correlation between D4A levels with clinical response will be performed by univariate and multivariate analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.
Locations (1):
- Sociedade Beneficiante de Senhoras - Hospital Sirio Libanes, São Paulo, Brazil